CLINICAL TRIAL: NCT02169635
Title: Safety and Efficacy Study of Macular Buckle With A Three-armed Silicone Capsule to Support the Posterior Staphyloma in High Myopia.
Brief Title: Macular Buckle With Three-armed Silicone
Acronym: MBTAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Lu, Director, Fundus Disease Center of Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013meky013
Record Dates: First submitted 2014-06-17; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: High Myopia; Posterior Staphyloma
Keywords: macular buckle; high myopia; posterior staphyloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Macula buckle (Experimental): Macular buckle: perform episcleral macular buckle surgery using a three-armed silicone capsule to support the posterior staphyloma in high myopia.
  Interventions: Procedure: macular buckle

INTERVENTIONS:
Procedure: macular buckle — macular buckle with a three-armed silicone capsule

SUMMARY:
High myopia is characterized by prolonged axial length and posterior staphyloma, which result in choroid-retinal degeneration and vision decrease. At present, vitrectomy can lead to anatomical improvements, but an higher axial length and the presence of a sever posterior staphyloma remains to be the two most important risk factors for poor visual outcomes. For these reasons, a different surgical approach, including macular buckling, might be considered in those patients with extremely high degree of myopia, in order to counteract the traction exerted by the posterior staphyloma. Macular buckling with or without pars plana vitrectomy had been proved to be an effective way to resolve myopic staphyloma related foveoschisis, macular hole, and associated retinal detachment. In this study, we sought to investigate the safety and efficacy of a macular buckling technique using a three-armed silicone capsule to support the posterior staphyloma in high myopia.

DETAILED DESCRIPTION:
1. This study plans to recruit 11 participants with 6 months follow-up to assess the safety and efficacy of a newly designed macular buckle device;
2. The macular buckle device, surgical procedure, and participants registry had been reviewed and approved by Ethics committee of Zhongshan Ophthalmic Center;
3. Only those patients are diagnosed with severe posterior staphyloma are registered.
4. All participants are fully informed before register;
5. All the surgeries are performed by single qualified doctor (Lin Lu);
6. After operation, all participant could contact the researcher via telephone, and could be assessed for any surgical related complications. If there is severe complication happened, or any person that could not tolerant the macular buckle, the implanted device will be removed;
7. Specially assigned staff (Jinge Lu) is responsible for data collection, data management, adverse events reporting, and participant communication.

ELIGIBILITY:
Inclusion Criteria:

* high myopia over -8.0 Diopter
* axial length over 26.5 mm
* posterior staphyloma

Exclusion Criteria:

* single eye patients
* retinal detachment beyond macular area
* a history of posterior scleritis
* a history of Glaucoma
* active hemorrhage in the surgical eye
* active inflammation in the surgical eye
* any situation that might hinder the observation of macular

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
best corrected visual acuity | 6 months

SECONDARY OUTCOMES:
postoperative complications | 6 months
Optical coherence tomography | 6 months
  Using optical coherence tomography to observe the macular area postoperatively.

OTHER OUTCOMES:
intraocular pressure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lu, MD, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Parolini B, Frisina R, Pinackatt S, Mete M. A new L-shaped design of macular buckle to support a posterior staphyloma in high myopia. Retina. 2013 Jul-Aug;33(7):1466-70. doi: 10.1097/IAE.0b013e31828e69ea. No abstract available. PMID 23619638
- [Background] Ward B. Degenerative myopia: myopic macular schisis and the posterior pole buckle. Retina. 2013 Jan;33(1):224-31. doi: 10.1097/IAE.0b013e31826d3a93. No abstract available. PMID 23190923
- [Background] Devin F, Tsui I, Morin B, Duprat JP, Hubschman JP. T-shaped scleral buckle for macular detachments in high myopes. Retina. 2011 Jan;31(1):177-80. doi: 10.1097/IAE.0b013e3181fc7e73. No abstract available. PMID 21102364
- [Background] Ward B, Tarutta EP, Mayer MJ. The efficacy and safety of posterior pole buckles in the control of progressive high myopia. Eye (Lond). 2009 Dec;23(12):2169-74. doi: 10.1038/eye.2008.433. PMID 19229272
- [Background] Alkabes M, Pichi F, Nucci P, Massaro D, Dutra Medeiros M, Corcostegui B, Mateo C. Anatomical and visual outcomes in high myopic macular hole (HM-MH) without retinal detachment: a review. Graefes Arch Clin Exp Ophthalmol. 2014 Feb;252(2):191-9. doi: 10.1007/s00417-013-2555-5. Epub 2014 Jan 3. PMID 24384802